CLINICAL TRIAL: NCT05907070
Title: The Effect of Mandala Art and Value Clarification Based on Watson's Theory of Human Caring on the Anxiety and Mood of Parents of Children With Cancer
Brief Title: Mandala Art and Value Clarification With Parents of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Meltem Gürcan, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023.9
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries
Keywords: child; value clarification; parent; cancer; mandala; art therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mandala group (Experimental): Mandala drawing and coloring on paper
  Interventions: Other: Mandala group
- Value clarification group (Experimental): Value clarification by writing on paper
  Interventions: Other: Value clarification group
- Control group (No Intervention): Routine nursing care

INTERVENTIONS:
Other: Mandala group — Mandala group will participate in 2 sessions of individual mandala drawing art activity with the theme of 'Emotions' accompanied by classical or instrumental music. In each session, a mandala will be created.
  Arms: Mandala group
Other: Value clarification group — Value clarification groups will participate in the value clarification activity by writing 2 sessions individually with the theme of 'Emotions' accompanied by classical or instrumental music.
  Arms: Value clarification group

SUMMARY:
The research is planned to be conducted with a randomized controlled experimental study. In the research, it is aimed to determine the effect of mandala drawing art and value clarification application based on Watson Human Care Theory on the anxiety and mood of the parents of children with cancer.

DETAILED DESCRIPTION:
The population of the study consists of the parents of children diagnosed with cancer in the Akdeniz University Hospital Pediatric Hematology and Oncology Clinic. The sample of the study is three groups; intervention 1 group (n:25), intervention 2 group (n:25) and control group (n:25) will consist of a total of 75 parents. A closed envelope system with simple randomization will be used in sample selection.

Intervention 1 group will participate in 2 sessions of individual mandala drawing art activity with the theme of 'Emotions' accompanied by classical or instrumental music. In each session, a mandala will be created. Intervention 2 groups will participate in the value clarification activity by writing 2 sessions individually with the theme of 'Emotions' accompanied by classical or instrumental music. Personal Information Form, State Anxiety Inventory and Positive-Negative Affect Scale were administered to the intervention groups at the first meeting in order to collect pre-test data. To collect post-test data, the State Anxiety Inventory and the Positive-Negative Affect Scale were administered immediately after the second session. No intervention will be made to the control group, the same data collection tools were applied to the intervention groups.

In addition, Iin the second session, the parent was asked to interpret the colors and shapes in the mandala created by the parent and a face-to-face interview was held.

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to read, write, speak and understand Turkish
* Being the parent of a 0-17-year-old child diagnosed with cancer
* Staying in the hospital with child
* Being hospitalized for at least the second course of treatment of the child

Exclusion Criteria:

* Having a physical problem that may prevent you from drawing and typing a mandala and participating in value clarification
* Not being able to take a break from caring for their child and participate in individual activities
* Having the child in the terminal period
* Relapse disease of the child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Positive-Negative Affect Scale (PANAS) | pre-test
  The scale consists of 20 items, 10 of which are positive and 10 of which are negative, describing various emotions. The scale has 2 sub-dimensions: positive and negative affect.
Positive-Negative Affect Scale (PANAS) | 2 or 3 days after pre-test
  The scale consists of 20 items, 10 of which are positive and 10 of which are negative, describing various emotions. The scale has 2 sub-dimensions: positive and negative affect.
State Anxiety Inventory (STAI) | pre-test
  The State Anxiety Inventory is a 4-point Likert-type scale consisting of 20 items. According to the level of life of individuals; It is answered by marking one of the options such as (1) not at all, (2) a little, (3) a lot, (4) completely.
State Anxiety Inventory (STAI) | 2 or 3 days after pre-test
  The State Anxiety Inventory is a 4-point Likert-type scale consisting of 20 items. According to the level of life of individuals; It is answered by marking one of the options such as (1) not at all, (2) a little, (3) a lot, (4) completely.

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan ATAY TURAN, PhD, Study Director — Assistant Professor
Locations (1):
- Meltem Gürcan, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No